CLINICAL TRIAL: NCT06848634
Title: Impact of Equestrian Sports, CrossFit, and Gym Training on Pelvic Floor Health in Athletes and Non-Athletes: A Cross-Sectional Study
Brief Title: Impact of Equestrian Sports, CrossFit, and Gym Training on Pelvic Floor Health (PELFISPORT )
Acronym: PELFISPORT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Maria Blanco Diaz, Principal investigator, University of Oviedo
Other Study IDs: EQUIPELVIC-001
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Floor Dysfunction; Urinary Incontinence; Pelvic Organ Prolapse (POP); Chronic Pelvic Pain
Keywords: Urinary incontinence; Pelvic organ prolapse; Chronic pelvic pain; Equestrian sports; CrossFit; Gym training; Women's health; Physical activity
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Equestrian: Participants who have been practicing equestrian sports for more than 2 years and train at least twice per week.
  This group will be assessed for pelvic floor dysfunction and compared with other sports disciplines and non-athletes.
- CrossFit: Participants engaged in CrossFit for at least 2 years, training at least twice per week.
  The study will evaluate how high-intensity training affects pelvic floor health.
- Gym Group: Participants who train in a gym (cardio, weightlifting, or fitness classes) for at least 2 years, with a minimum frequency of twice per week.
  The study aims to assess the impact of different gym training modalities on pelvic health.
- Other Sports Group: Participants engaged in other sports (e.g., swimming, cycling, team sports) for at least 2 years, training at least twice per week.
  This group provides a broader comparison of pelvic floor health across different physical activities.
- Non-Athletes Group: Participants who do not engage in regular physical activity. This group serves as a baseline comparison to evaluate the potential impact of sports on pelvic floor health.

SUMMARY:
This observational cross-sectional study investigates the impact of equestrian sports, CrossFit, and gym training on pelvic floor health in both athletes and non-athletes. The study aims to determine whether specific sports are associated with a higher risk of pelvic floor dysfunction, including urinary incontinence, pelvic organ prolapse, and chronic pelvic pain.

Participants will complete an online survey that collects demographic information, sports participation details, and pelvic floor health symptoms. The survey includes standardized questionnaires to assess pelvic floor function. Data will be analyzed to compare the prevalence of pelvic floor issues among different sports and between athletes and non-athletes.

The study seeks to provide insights into how sports participation influences pelvic health and to raise awareness of pelvic floor dysfunction in both male and female athletes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older.
* Voluntary participation with signed informed consent.
* Completion of the online survey.
* For the sports groups (Equestrian, CrossFit, Gym, Other Sports):

  * Minimum 2 years of experience in the sport.
  * Minimum 2 training sessions per week.

Exclusion Criteria:

* Individuals under 18 years old.
* Participants who do not complete the survey.
* Individuals with neurological conditions affecting mobility.
* Individuals with mobility impairments unrelated to sports.
* Sports participants with less than 2 years of experience or training less than twice per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes adults aged 18 and older who voluntarily participate by completing an online survey on pelvic floor health and sports practice. The study targets both athletes (equestrian sports, CrossFit, gym training, and other sports) and non-athletes to compare the prevalence of pelvic floor dysfunction across different activity levels.
  Participants in the sports groups must have at least two years of experience in their respective sport and train at least twice per week. The survey is distributed via social media, sports federations, gyms, and CrossFit centers to ensure a diverse sample.
  The study aims to provide insights into the impact of sports participation on pelvic floor health and identify potential risk factors for dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Pelvic Floor Dysfunction Among Different Sports Groups | Baseline (At the time of survey completion (single assessment point))
  Percentage of participants reporting symptoms of pelvic floor dysfunction (urinary incontinence, prolapse, chronic pelvic pain) across different sports groups and non-athletes.

SECONDARY OUTCOMES:
Impact of Sports Frequency on Pelvic Floor Dysfunction | Baseline (At the time of survey completion (single assessment point))
  Correlation between training frequency (sessions per week) and severity of pelvic floor symptoms.
Effect of Childbirth History on Pelvic Floor Dysfunction checklist | Baseline (At the time of survey completion (single assessment point))
  Comparison of pelvic floor symptoms between women with and without childbirth history, including mode of delivery.
Perceived Impact of Menstrual Cycle on Athletic Performance | Baseline (At the time of survey completion (single assessment point))
  Self-reported impact of menstrual symptoms on sports performance, using a 0-10 scale.

IPD SHARING:
Plan to Share IPD: No